CLINICAL TRIAL: NCT00071292
Title: Mindfulness Meditation-Based Stress Reduction in Relieving Symptoms Associated With Rheumatoid Arthritis
Brief Title: Meditation-Based Stress Reduction in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: P50AT000084 (NIH); Pradhan, Elizabeth
Record Dates: First submitted 2003-10-17; First posted 2003-10-21 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; stress reduction; meditation; mindfulness; MBSR; mindfulness-based stress reduction; mind-body skills
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meditation

INTERVENTIONS:
Behavioral: stress reduction program
Behavioral: meditation

SUMMARY:
The purpose of this study is to determine whether a mindfulness meditation-based stress reduction program is useful in relieving symptoms associated with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of RA, with doctor's letter or doctors' bill with ICD code 714;
* 18 years of age or older;
* Able to read and write English;
* Able to attend 15 course sessions and questionnaire sessions at Kernan Hospital in Baltimore;
* Willing to practice skills for 45 minutes to 1 hour per day, 6 days a week;
* Stable on rheumatoid medications for at least one month.

Exclusion criteria:

* Major psychiatric illness (bipolar disorder, multiple personality disorder, etc.);
* Active alcoholism or drug dependency;
* Scheduled for major surgery during the study period;
* Enrolled in randomized clinical trial for rheumatoid arthritis during the study period;
* Planning to move out of the area in the next 12 months;
* Unwilling to be enrolled in a control group;
* Use of assistive device other than a cane;
* Serious health condition(s) that the investigator determines would make it difficult to complete the 6 month study;
* Diagnosis of fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-07; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, Principal Investigator — Director, Center for Integrative Medicine
Locations (1):
- University of Maryland School of Medicine - Kernan Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn J, Lipworth L, Burney R. The clinical use of mindfulness meditation for the self-regulation of chronic pain. J Behav Med. 1985 Jun;8(2):163-90. doi: 10.1007/BF00845519. PMID 3897551
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Miller JJ, Fletcher K, Kabat-Zinn J. Three-year follow-up and clinical implications of a mindfulness meditation-based stress reduction intervention in the treatment of anxiety disorders. Gen Hosp Psychiatry. 1995 May;17(3):192-200. doi: 10.1016/0163-8343(95)00025-m. PMID 7649463
- [Background] Kaplan KH, Goldenberg DL, Galvin-Nadeau M. The impact of a meditation-based stress reduction program on fibromyalgia. Gen Hosp Psychiatry. 1993 Sep;15(5):284-9. doi: 10.1016/0163-8343(93)90020-o. PMID 8307341